CLINICAL TRIAL: NCT00454207
Title: A Phase 3, Multi-Center, Open-Label Study to Assess Safety and Efficacy of Sildenafil Citrate 20 mg TID in Subjects With Pulmonary Arterial Hypertension
Brief Title: Open Label Study of Sildenafil in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481252; JapicCTI-070381
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension, PAH
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sildenafil citrate (UK-92,480) (Experimental): sildenafil citrate 20 mg TID
  Interventions: Drug: sildenafil citrate (UK-92,480)

INTERVENTIONS:
Drug: sildenafil citrate (UK-92,480) — sildenafil citrate (UK-92,480)

SUMMARY:
To assess the safety of sildenafil 20 mg TID orally given to Japanese pulmonary arterial hypertension patients (Part 1 and 2) To assess the efficacy after 12 weeks of treatment of sildenafil 20 mg TID orally given to Japanese pulmonary arterial hypertension patients (Part 1)

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 16 and over, and classified as having pulmonary arterial hypertension
* Subjects who meet the following conditions on right heart catheterization at screening or baseline: mean pulmonary arterial pressure of ≥ 25mmHg and pulmonary capillary wedge pressure of ≤ 15mmHg at rest
* Subjects whose baseline 6-Minute Walk test distance is >100 m and <450 m

Exclusion Criteria:

* Significant Hepatic and/or renal disorder
* Subjects with known hereditary degenerative retinal disorders (such as retinitis pigmentosa) or history of non-arteritic ischemic optic neuropathy (NAION)
* Subjects who are currently receiving nitrates or nitric oxide donors in any form, ritonavir, ketoconazole and itraconazole

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481252&StudyName=Open%20Label%20Study%20of%20Sildenafil%20in%20Patients%20with%20Pulmonary%20Arterial%20Hypertension%20%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight centers in Japan
Pre-assignment Details: Twenty-one pulmonary arterial hypertension patients who have never received sildenafil therapy entered the study from Part I period and could continue to study part II period. Twenty-three patients who were continuously using sildenafil entered the study from Part II period.
Groups:
- Sildenafil: Participant Who Entered the Study From Part I: Consists of participants who entered the study from Part I period in Week 0. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil: Participants Who Entered the Study From Part II: Consists of participants who newly entered the study from Part II period in Week 0. The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to subjects after approval for the indication of pulmonary arterial hypertension).
Period: Overall Study
Arm/Group | Sildenafil: Participant Who Entered the Study From Part I | Sildenafil: Participants Who Entered the Study From Part II
Started | 21 | 23
Completed | 17 (19 participants completed Part I period. 17 of 19 participants continued from part I into Part II.) | 21
Not Completed | 4 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil: Participant Who Entered the Study From Part I | Sildenafil: Participants Who Entered the Study From Part II | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Japan | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in the 6-minute Walk Distance From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：6-minute walk distance at Week 12 minus 6-minute walk distance at baseline. The 6-minute walk distance:total distance walked during the 6-minute walk test.
Time Frame: Baseline, Week 12
Population: Full Analysis Set, including participants who took at least one dose of study medication and had efficacy measurements at both baseline and post-baseline. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Sildenafil: Part I: Consists of participants who entered the study from Part I period in Week 0. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil: Part I
Number analyzed (Participants) | 20
meters | 84.2 (74.9)

2. Primary Outcome: Change in the Mean Pulmonary Arterial Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change:Mean pulmonary arterial pressure at Week 12 minus mean pulmonary arterial pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sildenafil:Part I: Consists of participants who entered the study from Part I period in Week 0. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -4.7 (8.2)

3. Primary Outcome: Change in the Pulmonary Vascular Resistance From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Pulmonary vascular resistance at Week 12 minus pulmonary vascular resistance at baseline
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dyne·second/centimeter^5
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
dyne·second/centimeter^5 | -246.49 (301.17)

4. Secondary Outcome: Change in the 6-minute Walk Distance From Baseline at Week 8 in Participants Who Entered the Study From Part I
Description: Change：6-minute walk distance at Week 8 minus 6-minute walk distance at baseline.
  The 6-minute walk distance:Total distance walked during the 6- minute walk test.
Time Frame: Baseline, Week 8
Population: Full Analysis Set, including participants who took at least one dose of study medication and had efficacy measurements at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 19
meters | 87.5 (75.3)

5. Secondary Outcome: Change in the Systolic Pulmonary Arterial Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Systolic pulmonary arterial pressure at Week 12 minus Systolic pulmonary arterial pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -3.4 (13.4)

6. Secondary Outcome: Change in the Diastolic Pulmonary Arterial Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Diastolic pulmonary arterial pressure at Week 12 minus diastolic pulmonary arterial pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -3.2 (8.3)

7. Secondary Outcome: Change in the Systolic Systemic Blood Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Systolic systemic blood pressure at Week 12 minus systolic systemic blood pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | 0.7 (16.5)

8. Secondary Outcome: Change in the Diastolic Systemic Blood Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Diastolic systemic blood pressure at Week 12 minus diastolic systemic blood pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -3.1 (9.0)

9. Secondary Outcome: Change in the Mean Systemic Blood Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Mean systemic blood pressure:diastolic blood pressure+(systolic blood pressure-diastolic blood pressure)/3.
  Change：Mean systemic blood pressure at Week 12 minus mean systemic blood pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -0.9 (12.9)

10. Primary Outcome: Change in the Cardiac Output From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Cardiac output at Week 12 minus cardiac output at baseline
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter/minute
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
liter/minute | 0.556 (1.000)

11. Secondary Outcome: Change in the Pulmonary Capillary Wedge Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Pulmonary capillary wedge pressure at Week 12 minus pulmonary capillary wedge pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | 0.68 (3.14)

12. Secondary Outcome: Change in the Right Atrial Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Right atrial pressure at Week 12 minus right atrial pressure at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -0.3 (4.4)

13. Secondary Outcome: Change in the Cardiac Index From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Cardiac index at Week 12 minus cardiac index at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter/minute/meter^2
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
liter/minute/meter^2 | 0.32 (0.62)

14. Secondary Outcome: Change in the Heart Rate From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Heart rate at Week 12 minus heart rate at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
beats/minute | -4.14 (7.45)

15. Secondary Outcome: Change in the Pulmonary Vascular Resistance Index From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change:Pulmonary vascular resistance index at Week 12 minus pulmonary vascular resistance index at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dyne*second/centimeter^5/meter^2
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
dyne*second/centimeter^5/meter^2 | -382.00 (491.80)

16. Secondary Outcome: Change in the Systemic Vascular Resistance From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Systemic vascular resistance at Week 12 minus systemic vascular resistance at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dyne*second/centimeter^5
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
dyne*second/centimeter^5 | -265.77 (785.52)

17. Secondary Outcome: Change in the Systemic Vascular Resistance Index From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Systemic vascular resistance index at Week 12 minus systemic vascular resistance index at baseline.
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dyne*second/centimeter^5/meter^2
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
dyne*second/centimeter^5/meter^2 | -409.89 (1271.30)

18. Secondary Outcome: Change in the Mixed Venous Oxygen Saturation From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Mixed venous oxygen saturation at Week 12 minus mixed venous oxygen saturation at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
percent saturation | 2.91 (9.05)

19. Secondary Outcome: Change in the Arterial Oxygen Saturation From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Arterial oxygen saturation at Week 12 minus arterial oxygen saturation at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
percent saturation | 0.440 (5.437)

20. Secondary Outcome: Change in the Arterial Oxygen Partial Pressure From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Arterial oxygen partial pressure at Week 12 minus arterial oxygen partial pressure at baseline.
Time Frame: baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
mmHg | -2.02 (11.17)

21. Secondary Outcome: Change in the Partial Pressure of Mixed Venous Oxygen From Baseline at Week 12 in Participants Who Entered the Study From Part I
Description: Change：Partial pressure of mixed venous oxygen at Week 12 minus partial pressure of mixed venous oxygen at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 19
mmHg | 0.57 (4.35)

22. Secondary Outcome: Changes in the World Health Organization (WHO) Functional Class of Pulmonary Arterial Hypertension From Baseline at Weeks 12 in Participants Who Entered the Study From Part I
Description: The cross-tabulation table on the WHO functional classes of pulmonary arterial hypertension at baseline and Week 12. The WHO functional classes of pulmonary arterial hypertension:Class I (pulmonary arterial hypertension patients with no limitation in physical activity) to Class IV (pulmonary arterial hypertension patients who can not perform a physical activity without any symptoms).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Sildenafil:Part I , Functional Class at Baseline: I: Consists of participants who entered the study from Part I period in Week 0, and whose WHO functional class at baseline were I. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil:Part I, Functional Class at Baseline: II: Consists of participants who entered the study from Part I period in Week 0, and whose WHO functional class at baseline were II. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil, Part I, Functional Class at Baseline: III: Consists of participants who entered the study from Part I period in Week 0, and whose WHO functional class at baseline were III. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil, Part I, Functional Class at Baseline:IV: Consists of participants who entered the study from Part I period in Week 0, and whose WHO functional class at baseline were IV. The participants were treated with sildenafil 20 mg three times a day orally in Part I period (12 weeks) and Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Part I , Functional Class at Baseline: I | Sildenafil:Part I, Functional Class at Baseline: II | Sildenafil, Part I, Functional Class at Baseline: III | Sildenafil, Part I, Functional Class at Baseline:IV
Number analyzed (Participants) | 0 | 7 | 13 | 0
participants
  Functional class at Week 12:I |  | 0 | 1 |
  Functional class at Week 12:II |  | 6 | 5 |
  Functional class at Week 12:III |  | 1 | 7 |
  Functional class at Week 12:IV |  | 0 | 0 |

23. Secondary Outcome: Changes in the BORG Dyspnoea Score From Baseline at Week 8 and Week 12 in Participants Who Entered the Study From Part I
Description: Change：BORG dyspnoea score at Week 8 and Week 12 minus BORG dyspnoea score at baseline. BORG dyspnoea score:Scale 0 (no breathlessness at all) to 10 (maximum). The score reflected the maximum degree of dyspnoea that the participants experienced at any time during the 6-minute walk distance.
Time Frame: Baseline, Week 8, Week 12
Population: Full Analysis Set, including participants who took at least one dose of study medication and had efficacy measurements at both baseline and post-baseline. Last observation carried forward (Week 12).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
scores on a scale
  Week 8 (n=19, 0) | -0.84 (1.89)
  Week 12 (n=20, 6) | -0.95 (1.94)

24. Secondary Outcome: Changes in the the Plasma Brain Natriuretic Peptide Level From Baseline at Week 4, Week 8 and Week 12 in Participants Who Entered the Study From Part I
Description: Change：Plasma brain natriuretic peptide level at Week 4, Week 8 and Week 12 minus plasma brain natriuretic peptide level at baseline
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Sildenafil:Part I
Number analyzed (Participants) | 20
picograms/milliliter
  Week 4 (n=20, 0) | -78.00 (166.41)
  Week 8 (n=19, 0) | -88.25 (178.39)
  Week 12 (n=20, 7) | -61.82 (209.96)

25. Secondary Outcome: Change in the 6-minute Walk Distance From Baseline at Week 12 in Participants Who Newly Entered the Study From Part II
Description: Change：6-minute walk distance at Week 12 minus 6-minute walk distance at baseline. The 6-minute walk distance:Total distance walked during the 6- minute walk test.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Sildenafil:Part II: Consists of participants who newly entered the study from Part II period in Week 0 and had been receiving sildenafil at doses higher than 60 mg/day before the start of this study. The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Part II
Number analyzed (Participants) | 7
meters | -23.5 (34.1)

26. Secondary Outcome: Change in the World Health Organization (WHO) Functional Class From Baseline at Week 12 in Participants Who Newly Entered the Study From Part II
Description: as for outcome 22
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Sildenafil:Part II, Functional Class at Baseline: I: Consists of participants who newly entered the study from Part II period in Week 0, and whose WHO functional class at baseline were I. The participants had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil:Part II, Functional Class at Baseline: II: Consists of participants who newly entered the study from Part II period in Week 0, and whose who functional class at baseline were II. The participants had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil: Part II, Functional Class at Baseline: III: Consists of participants who newly entered the study from Part II period in Week 0, and whose WHO functional class at baseline were III. The participants had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
- Sildenafil: Part II, Functional Class at Baseline: IV: Consists of participants who newly entered the study from Part II period in Week 0, and whose WHO functional class at baseline were IV. The participants had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Part II, Functional Class at Baseline: I | Sildenafil:Part II, Functional Class at Baseline: II | Sildenafil: Part II, Functional Class at Baseline: III | Sildenafil: Part II, Functional Class at Baseline: IV
Number analyzed (Participants) | 1 | 6 | 0 | 0
participants
  Functional class at Week 12: I | 1 | 0 |  |
  Functional class at Week 12: II | 0 | 5 |  |
  Functional class at Week 12: III | 0 | 1 |  |
  Functional class at Week 12: IV | 0 | 0 |  |

27. Secondary Outcome: Changes in the BORG Dyspnoea Score From Baseline at Week 12 in Participants Who Newly Entered the Study From Part II
Description: Change：BORG dyspnoea score at Week 12 minus BORG dyspnoea score at baseline. BORG dyspnoea score:Scale 0 (no breathlessness at all) to 10 (maximum). The score reflected the maximum degree of dyspnoea that the participants experienced at any time during the 6-minute walk distance.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Sildenafil: Part II: Consists of participants who newly entered the study from Part II period in Week 0 and had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil: Part II
Number analyzed (Participants) | 6
scores on a scale | 0.33 (1.21)

28. Secondary Outcome: Changes in the the Plasma Brain Natriuretic Peptide Level From Baseline at Week 12 in Participants Who Newly Enterd the Study From Part II
Description: Change：Plasma brain natriuretic peptide level at Week 12 minus plasma brain natriuretic peptide level at baseline
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Groups:
- Sildenafil:Part II: Consists of participants who newly entered the study from Part II period in Week 0 and had been receiving sildenafil at doses higher than 60 mg/day before the start of this study.The participants were treated with sildenafil 20 mg three times a day orally in Part II period (long-term treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Part II
Number analyzed (Participants) | 7
picograms/milliliter | 15.91 (55.94)

29. Secondary Outcome: Maximum Plasma Concentrations (Cmax) of Sildenafil and Sildenafil's Metabolite, UK-103,320
Description: Maximum plasma concentrations was calculated from the observed value of plasma concentrations in each participant
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours after dosing
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Groups:
- Sildenafil:Pharmacokinetic Analysis Participant: Consists of participants who received sildenafil monotherapy, without administration of other treatment drugs for pulmonary arterial hypertension, in Part I or II, and satisfied the inclusion criteria for pharmacokinetics evaluation without violating the exclusion criteria. The participants were treated with sildenafil 20 mg three times a day orally in Part I period(12 weeks) and Part II period (longterm treatment period, until a proper system was established to provide sildenafil to participants after approval for the indication of pulmonary arterial hypertension).
Arm/Group | Sildenafil:Pharmacokinetic Analysis Participant
Number analyzed (Participants) | 9
nanograms/milliliter
  Sildenafil | 164.88 (74.78)
  Sildenafil's Metabolite, UK-103,320 | 87.27 (30.67)

30. Secondary Outcome: Time to First Occurrence of Maximum Plasma Concentrations (Tmax) of Sildenafil and Sildenafil's Metabolite, UK-103,320
Description: Time to first occurrence of maximum plasma concentrations were calculated from the observed value of plasma concentrations in each participant.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours after dosing
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sildenafil:Pharmacokinetic Analysis Participant
Number analyzed (Participants) | 9
hours
  Sildenafil | 1.102 (0.499)
  Sildenafil's Metabolite, UK-103,320 | 1.611 (1.024)

31. Secondary Outcome: The Area Under the Curve (AUC) From Time 0 to Time 8 Hour of Sildenafil and Sildenafil's Metabolite, UK-103,320
Description: The area under the curve from time 0 to time 8 hour was calculated from area under the curve in each perticipant on the date of blood sampling using the linear/log trapezoidal rule
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours after dosing
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter
Arm/Group | Sildenafil:Pharmacokinetic Analysis Participant
Number analyzed (Participants) | 9
nanogram*hour/milliliter
  Sildenafil | 545.14 (294.88)
  Sildenafil's Metabolite, UK-103,320 | 365.85 (186.55)

32. Secondary Outcome: The Average Plasma Concentration (Css,av) of Sildenafil at Steady State
Description: The average plasma concentration of sildenafil at steady state was calculated from the area under the curve from time 0 to 8 hour/dosing interval (8 hours).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours after dosing
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Sildenafil:Pharmacokinetic Analysis Participant
Number analyzed (Participants) | 9
nanograms/milliliter | 68.14 (36.86)

33. Secondary Outcome: The Average Plasma Trough Concentration (Ctrough) of Sildenafil
Description: The average plasma trough concentration of sildenafil was calculated from the observed value before administration of the drug in each participants.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours after dosing
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Sildenafil:Pharmacokinetic Analysis Participant
Number analyzed (Participants) | 9
nanograms/milliliter | 19.608 (12.438)

34. Secondary Outcome: Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: The total number of participants with laboratory test abnormalities without regard to baseline abnormality.
Time Frame: Baseline up to 1.3 years
Population: All subjects who received at least one dose of the study medication and had any evaluable laboratory test data after treatment.
Measure: Number; unit: participants
Groups:
- Sildenafil: Part I and Part II: Consists of participants who entered the study from Part I period plus participants who entered the study from Part II period.
Arm/Group | Sildenafil: Part I and Part II
Number analyzed (Participants) | 43
participants | 35

ADVERSE EVENTS:
Arm/Group | Sildenafil: Part I and Part II
Serious Adverse Events (participants affected / at risk) | 7/44
Other Adverse Events (participants affected / at risk) | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil: Part I and Part II (N=44)
Cardiac failure (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Scleroderma renal crisis (Renal and urinary disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil: Part I and Part II (N=44)
Diarrhoea (Gastrointestinal disorders) | 4
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 17
Fall (Injury, poisoning and procedural complications) | 4
Platelet count decreased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Flushing (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.